CLINICAL TRIAL: NCT00002364
Title: An Exploratory Study of the Antiretroviral Activity of 1592U89 When Administered in Combination With Other Specific Nucleoside Reverse Transcriptase Inhibitors (NRTIs) in NRTI Experienced Patients
Brief Title: A Study of 1592U89 Combined With Other Anti-HIV Drugs in Patients Who Have Taken Anti-HIV Drugs
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Glaxo Wellcome (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 238C; CNAA 2003
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1997-04

CONDITIONS: HIV Infections
Keywords: Drug Therapy, Combination; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Antiviral Agents
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — abacavir

INTERVENTIONS:
Drug: Abacavir sulfate

SUMMARY:
To obtain preliminary evidence of antiretroviral activity of 1592U89 when administered in combination with other specific NRTI agents in NRTI experienced patients and to assess the safety and tolerance of multiple oral doses of 1592U89 when administered in combination with specific marketed NRTIs.

DETAILED DESCRIPTION:
Patients will all receive oral doses of 1592U89 in combination with protocol specific current antiretroviral therapy. The treatment groups will be assigned based on each subject's previous NRTI experience.

The study medication is self administered and all evaluations will be performed on an outpatient basis. Patients will be seen at day 0 and weeks 2, 4, 12, 16, 20 and 24.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* CD4+ cell count >= 100 /mm3.
* Plasma HIV RNA >= 30,000 copies/ml.
* Study participants may be recruited from all clinical categories, provided they do not meet any of the exclusion criteria.
* Parent or legal guardian to sign written, informed consent for patients under the age of 18.

Exclusion Criteria

Co-existing Condition:

Patients with any of the following symptoms or conditions are excluded:

* Patients with active or ongoing AIDS-defining opportunistic infection or disease. NOTE:
* For this study, a CD4+ cell count <= 200 cells/mm3 in the absence of any other AIDS defining indicator condition is not considered an AIDS defining event.
* Malabsorption syndrome or other gastrointestinal dysfunction that might interfere with drug absorption.
* Patients with life threatening infection or other serious medical conditions whose participation may compromise patient safety.

Concurrent Medication:

Excluded:

* Treatment with cytotoxic chemotherapeutic agents within the 24 weeks of the study.
* Patients receiving other investigational drugs.
* Foscarnet therapy or therapy with other agents with documented activity against HIV in vitro.
* Treatment with immunomodulators.
* Patients on methadone.

Concurrent Treatment:

Excluded:

* Treatment with radiation therapy within the 24 weeks of the study. NOTE:
* Localized radiation therapy may be permitted following consultation with the sponsor.

Patients with any of the following prior conditions are excluded:

* Subjects with a history of lymphoma.
* Subjects with a history of clinically apparent pancreatitis or hepatitis within the last 6 months.

Prior Medication:

Excluded:

* Treatment with any antiretroviral therapy with NRTIs (alone or in combination) other than those defined for each treatment group.
* Treatment with any non-nucleoside RT inhibitors or protease inhibitors.
* Treatment with cytotoxic chemotherapeutic agents within 1 month prior to study entry.
* Investigational HIV vaccine within the past 3 months.
* Immunomodulating agents such as systematic corticosteroids, interleukins, thalidomide, anticytokine agents, anti-oxidants or interferons within 1 month of study entry.

Prior Treatment:

Excluded:

* Treatment with radiation therapy within 1 month of entry.

Risk Behavior:

Excluded:

Patients with current alcohol or illicit drug use that, in the opinion of the principal investigator, may interfere with the patient's ability to comply with the study protocol.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Marin County Specialty Clinic, Greenbrae, California
  - Kraus Med Partners, Los Angeles, California
  - ViRx Inc, San Francisco, California
  - IDC Research Initiative, Altamonte Springs, Florida
  - North Broward Hosp District, Fort Lauderdale, Florida
  - AIDS Research Consortium of Atlanta, Atlanta, Georgia
  - Univ of Kentucky Med Ctr, Lexington, Kentucky
  - Beth Israel Med Ctr, New York, New York